CLINICAL TRIAL: NCT02562911
Title: Epidemiological Study of the Progress of Puberty in Girls Followed for Cystic Fibrosis
Brief Title: Puberty in Girls Followed for Cystic Fibrosis
Acronym: EPIMUCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 12 485 03
Record Dates: First submitted 2015-08-24; First posted 2015-09-29 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; menstrual cycle; puberty
MeSH Terms: conditions — Cystic Fibrosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Data collection — * Clinical examination
  * Complete pelvic ultrasound abdominal ultrasound
  * Bone age: X-ray
  * biological examination
  * Lung function assessed by the Maximum Volume Expired
  * Brasfield radiological score (if available)

SUMMARY:
In the general population, age of puberty, and age of menarche in girls, are closely correlated with those of their mother. The severity of chronic disease has an impact on the stature, the weight gain and the onset of puberty: age of menarche is even later that chronic illness is serious. Cystic fibrosis is one of the major chronic diseases of children.

Neonatal screening is organized since 2002, most girls with cystic fibrosis therefore currently have a very specialized and early care. Older patients were diagnosed during childhood. The optimization of the nutritional and respiratory management has allowed over the past two decades a significant improvement in the survival of these patients. Most young people reach adulthood, puberty and reproductive desire are a crucial issue in the care of these young adults.

In literature, it is often noted an age of menarche delayed an average of 2 years compared to the general population, but correlated with the age of menstruation from the mothers.

The factors involved in the conduct of cycles in the girl followed for cystic fibrosis are poorly known and there are few data on the characteristics of cycles. The menstrual irregularity and amenorrhoea episodes concern nearly half of women.

On the pathophysiological level, studies in animals show that there is a direct effect of CFTR (Cystic Fibrosis Transmembrane Regulator) on the hypothalamic pituitary gonadal and reproductive capacity in mice.

The literature data on the pubertal development, fertility and hormonal profile of these girls are for studies with low numbers and are very old. There is to date no French cohort study on this topic.

The study is a multicenter cross-sectional descriptive study for pubertal and gynecological characteristics in girls followed annually in the reference centers Cystic Fibrosis two inter-region.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with cystic fibrosis
* Girl aged 8 years of age, adolescents and young adults, had period or not,
* visit the Reference and Competence Center of Cystic Fibrosis.
* Affiliated to a social security scheme

Exclusion Criteria:

* Lack of consent of the legal representative or the relevant patient.
* Patient majoring in legal disability or minor patient whose legal representative is legal disability

Min Age: 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Girl aged 8 years of age, adolescents and young adults, had period or not, visit the Reference and Competence Center of Cystic Fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The age of menarche in girls followed for cystic fibrosis in France | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Catherine PIENKOWSKI, MD, Principal Investigator — University Hospital, Toulouse
Locations (7):
- France (7):
  - CHU Besançon St Jacques, Besançon
  - Hôpital des Enfants-Pellegrin, Bordeaux
  - Hôpital d'Enfants, Dijon
  - Canton- Hôpitaux de Brabois, Nancy
  - American Memorial Hospital, Reims
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital des enfants Purpan, Toulouse